CLINICAL TRIAL: NCT07335965
Title: Study of the Clinical, Microbiological, and Epidemiological Characteristics of Recurrent Imported Borreliosis Confirmed by the Borrelia National Reference Center
Brief Title: Study of the Clinical, Microbiological and Epidemiological Characteristics of Recurrent Imported Borreliosis Confirmed by the CNR Borrelia
Acronym: BORRECUR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9541
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Borrelia Recurrentis Infection
Keywords: Borrelia Infections; Borrelia Recurrentis Infection
MeSH Terms: conditions — Relapsing Fever; Borrelia Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recurrent borreliosis (RB) is a bacterial infection transmitted by ticks or lice. These infections occur in both temperate and tropical regions, but are rare in Australia and Antarctica. Due to climate change, the areas inhabited by the vectors of these infections are shifting, and the number of at-risk regions has significantly increased in recent years. More than twenty RB species have been described, responsible for variable clinical manifestations including fever, myalgia, digestive disorders, and sometimes neurological symptoms. Tick-borne RB represents a major public health problem, particularly in Africa. Mortality from these infections ranges from 5% to 10%. In recent years, diagnostic techniques have evolved. Microscopic diagnosis was initially the gold standard but had only moderate sensitivity and exhibited inter-operator variability. The advent of molecular biology now allows for increased sensitivity with excellent specificity and also enables the identification of the causative species.

A few cases have been described in France, consisting mainly of case reports. Therefore, this study will provide a comparative description, within a series, of cases diagnosed in France: symptoms, patients' countries of origin, Borrelia species, diagnostic techniques, management, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult subject
* Having presented (from January 1, 2013, to January 1, 2025) with recurrent imported borreliosis, the diagnosis of which was confirmed by the CNR Borrelia in Strasbourg

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Minor or adult subject having presented (from January 1, 2013, to January 1, 2025) with recurrent imported borreliosis, the diagnosis of which was confirmed by the CNR Borrelia in Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Clinical and biological description of cases of recurrent imported borreliosis | Up to 12 years
  This study does not include any evaluation, but simply describes cases diagnosed in France: symptoms, patients' countries of origin, Borrelia species, diagnostic techniques, and treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire de Bactériologie - CHU de Strasbourg - France, Strasbourg, France